CLINICAL TRIAL: NCT01422382
Title: Drug-Drug Interaction Study to Assess the Effects of Steady-State Cardizem LA (Diltiazem Hydrochloride) and Steady-State Pitavastatin on Their Respective Pharmacokinetics in Healthy Adult Volunteers
Brief Title: Drug-Drug Interaction of Cardizem LA (Diltiazem Hydrochloride) on Pitavastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: NK-104-4.07US
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — pitavastatin; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental): There was 1 treatment period, with each subject receiving a once-daily dose of pitavastatin 4 mg on Days 1 through 5 and on Days 11 through 15 and a once-daily dose of diltiazem 240 mg on Days 6 through 15
  Interventions: Drug: Pitavastatin (NK-104); Drug: Diltiazem (Cardizem LA) 240 mg QD

INTERVENTIONS:
Drug: Pitavastatin (NK-104) — pitavastatin (NK-104) 4 mg once daily (QD)
  Other Names: Livalo
Drug: Diltiazem (Cardizem LA) 240 mg QD — Diltiazem (Cardizem LA) 240 mg QD

SUMMARY:
This is a Phase 4, single-center, open-label, fixed-sequence, multiple-dose, 2-way drug-drug interaction study.

DETAILED DESCRIPTION:
Each subject will qualify for entry into the study not more than 30 days prior to admission into the clinical unit. Subjects will check into the clinical unit on Day -1 for baseline assessments. During the treatment period, each subject will receive a once-daily dose of pitavastatin 4 mg on Days 1 through 5 and on Days 11 through 15 and a once-daily dose of diltiazem 240 mg on Days 6 through 15. Subjects will fast overnight for at least 8 hours before dosing and will remain fasted until 4 hours after dosing on the morning of Days 5, 10, and 15.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteer aged 18 to 45 years, inclusive.
* Subject has a body mass index of 18 to 30 kg/m2, inclusive.
* Subject has normal hematology, serum chemistry, and urinalysis test results.
* Subject is able and willing to abstain from alcohol, grapefruit-containing foods or beverages, caffeine, or caffeine-containing products, St John's wort, and herbal supplements for 4 days before Day 1 and until after completion of this study.
* Subject is a nonsmoker or has quit smoking at least 6 months before the first dose of study drug and until after study completion.

Exclusion Criteria:

* Subject has had any surgery of the gastrointestinal tract likely to affect drug absorption, distribution, metabolism, or excretion.
* Subject has had a previous allergy or intolerance to treatment with pitavastatin, diltiazem, or any drugs in these classes.
* Subject has a history of drug or alcohol abuse.
* Subject has had a clinically significant illness within 4 weeks before the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Morgan, MD, FACS, Study Director — Kowa Research Institute, Inc.
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1st Subject Enrolled 05 May 2011, Last Subject Completed 12 July 2011 at PPD Inc. 7551 Metro Center Drive Suite 200 Austin, TX 78744
Groups:
- All Subjects: All randomized subjects.
Period: NK-104 4mg Once Daily (QD)
Arm/Group | All Subjects
Started | 28
Completed | 28
Not Completed | 0
Period: Diltiazem 240 mg QD
Arm/Group | All Subjects
Started | 28
Completed | 28
Not Completed | 0
Period: NK-104 4mg QD and Diltiazem 240 mg QD
Arm/Group | All Subjects
Started | 28
Completed | 27
Not Completed | 1
Not completed — personal reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.2 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: NK-104 AUC
Time Frame: 15 Days
Population: All subjects with measurable pharmacokinetic (PK) values
Measure: Mean (Standard Deviation); unit: ng * h/mL
Arm/Group | All Subjects
Number analyzed (Participants) | 26
ng * h/mL | 208.92 (86.54)

2. Secondary Outcome: Number of Participants With at Least One Adverse Event.
Time Frame: 24 Days
Measure: Number; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 28
Participants | 12

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 12/28
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=28)
Headache (Nervous system disorders) | 5
Presyncope (Nervous system disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
May not publish.